CLINICAL TRIAL: NCT05655429
Title: Physical Therapy vs Arthroscopic Partial Meniscectomy on the Knee Function of Metabolic Syndrome Patients With Degenerative Meniscus Lesions
Brief Title: Physical Therapy vs Arthroscopic Partial Meniscectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ShenzhenPH meniscus001
Record Dates: First submitted 2022-12-02; First posted 2022-12-19 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Knee Medial Meniscus Tears
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- physical therapy (Experimental): Physical therapy mainly include aerobic exercises and resistance exercise, flexibility exercises about 150 minutes for ≥2 d/week for 6 months.
  Interventions: Procedure: physical therapy
- arthroscopic partial meniscectomy (Active Comparator): The torn meniscus and unstable part were removed with arthroscopic instruments.
  Interventions: Procedure: arthroscopic partial meniscectomy

INTERVENTIONS:
Procedure: physical therapy — The exercise intervention included aerobic exercises and resistance exercise, flexibility exercises about 150 minutes for ≥2 day per week.
  Arms: physical therapy
Procedure: arthroscopic partial meniscectomy — Arthroscopic partial meniscectomy surgery procedure
  Arms: arthroscopic partial meniscectomy

SUMMARY:
The purpose was to assess knee function outcomes between physical therapy and arthroscopic partial menisectomy(APM) for Metabolic syndrome(MetS) patients with degenerative meniscus lesions(DMLs) during 12 month follow up.

DETAILED DESCRIPTION:
Metabolic syndrome were diagnosed with abdominal obesity, insulin resistance with or without glucose intolerance, dyslipidemia or elevated blood pressure and widely prevalence all around the world.MetS patients were always correlated with knee osteoarthritis or cartilage volume loss. For MetS patients with DMLs, whether physical therapy was non-inferior to APM in knee function and MetS components was unknown.

ELIGIBILITY:
Inclusion Criteria:

* Must be age between 35 and 70 years old;

  * Clinical diagnosis of metabolic syndrome;
  * Clinical diagnosis of degenerative meniscus lesions;
  * Patients who has knee pain history
  * Knee symptoms consistent with DMLs verified on MRI
  * eligible for arthroscopic partial meniscectomy surgery by the examining orthopedic surgeons.

Exclusion Criteria:

* Must be able to have no acute knee injury such as car crash or acute sports injury;

  * Must be able to have no knee surgeries history;
  * Must be able to have no rheumatoid arthritis or serious knee osteoarthritis with deformity;
  * Must be able to have no contraindications to MRI;
  * Must be able to have no severe cardiopulmonary disease;
  * Must be able to have no musculoskeletal or neuromuscular impairments ;
  * Must be able to have good visual, hearing, or cognitive;

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-01-15 (Actual); Primary Completion 2023-08-02 (Estimated); Study Completion 2023-08-10 (Estimated)

PRIMARY OUTCOMES:
the Knee Injury and Osteoarthritis Outcome Score (KOOS) change | change from baseline up to 12 months
  The Knee injury and Osteoarthritis Outcome Score (KOOS) holds five subscales including: Pain (9 items); other Symptoms (7 items); Activities of Daily Living (ADL, 17 items); Sport and Recreation function (Sport/Rec, 5 items); and knee-related Quality of Life (QoL, 4 items). Each subscale is scored separately from zero (extreme knee problems) to 100 (no knee problems)
the International Knee Documentation Committee Subjective Knee Evaluation Form (IKDC Score) change | change from baseline up to 12 months
  The International Knee Documentation Committee Subjective Knee Evaluation Form (IKDC) score questionnaire contains 18 items (7 items for symptoms, 1 item for sport activity, 9 items for daily activities, and 1 item for current knee function.) The total score is transformed to a value on a scale of 0 to 100, with 100 representing the highest knee function and 0 is the worst.
waist circumstance change | change from baseline up to 12 months
  waist circumstance (cm)
systolic blood pressure change | change from baseline up to 12 months
  systolic blood pressure /mmHg
diastolic blood pressure change | change from baseline up to 12 months
  diastolic blood pressure/mmHg
serum total cholesterol (TC) change | change from baseline up to 12 months
  serum total cholesterol (TC) (mmol/L)
serum triglycerides (TG) change | change from baseline up to 12 months
  serum triglycerides (TG) (mmol/L)
low-density lipoprotein cholesterol (LDL-C) change | change from baseline up to 12 months
  serum low-density lipoprotein cholesterol (LDL-C) (mmol/L)
high-density lipoprotein cholesterol (HDL-C) change | change from baseline up to 12 months
  serum high-density lipoprotein cholesterol (HDL-C) (mmol/L)
fast blood glucose(FBG) change | change from baseline up to 12 months
  serum fast blood glucose(FBG) (mmol/L)
Body mass index change | change from baseline up to 12 months
  Body mass index(BMI) weight/height square (kg/㎡)
Kellgren-Lawrence (K/L) grade change | change from baseline up to 12 months
  Kellgren-Lawrence (K/L) grade

SECONDARY OUTCOMES:
pain score change | change from baseline up to 12 months
  The minimum is 0 points, the maximum is 4 points, from extreme knee problems to no knee problems. After the score of each part is calculated separately, it is converted into a percentage score by the conversion formula.
symptoms score change | change from baseline up to 12 months
  The minimum is 0 points, the maximum is 4 points, from extreme knee problems to no knee problems. After the score of each part is calculated separately, it is converted into a percentage score by the conversion formula.
activities of daily living score change | change from baseline up to 12 months
  The minimum is 0 points, the maximum is 4 points, from extreme knee problems to no knee problems. After the score of each part is calculated separately, it is converted into a percentage score by the conversion formula
function in sport and recreation score change | change from baseline up to 12 months
  The minimum is 0 points, the maximum is 4 points, from extreme knee problems to no knee problems. After the score of each part is calculated separately, it is converted into a percentage score by the conversion formula
knee related quality of life score change | change from baseline up to 12 months
  The minimum is 0 points, the maximum is 4 points, from extreme knee problems to no knee problems. After the score of each part is calculated separately, it is converted into a percentage score by the conversion formula

CONTACTS AND LOCATIONS:
Locations (1):
- Shenzhen People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No